CLINICAL TRIAL: NCT06034704
Title: Investigation of the Effect of Plantar Fascia Release With Magnetic Fascia Ball on Hamstring and Lumbar Spine Flexibility
Brief Title: Plantar Fascia Release With Magnetic Fascia Ball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-OOP-1
Record Dates: First submitted 2023-08-30; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Flexibility; Muscle Tightness
Keywords: Massage; Hamstring Muscles; Magnets; Lumbar Fascia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Fascial Ball (Experimental): In the experimental group, a fascial ball made of cork containing 3 magnets of 0.15 tesla was used. The magnetic fascia ball diameter is 6 centimetres.
  Interventions: Other: Plantar fascia self massage with a magnetic fascia ball
- Non-Magnetic Fascial Ball (Placebo Comparator): In the placebo group, a fascial ball made of cork without magnets. The non-magnetic fascia ball diameter is 6 centimetres.
  Interventions: Other: Plantar fascia self massage with a non-magnetic fascia ball

INTERVENTIONS:
Other: Plantar fascia self massage with a magnetic fascia ball — Participants were asked to roll the magnetic fascia ball on the sole of each foot for 3 minutes each, from the metatarsal heads towards the heel, concentrating on the medial longitudinal arch. Participants were informed that more intense pressure would be more beneficial and were asked to apply pressure in a way that would not cause pain.
  Arms: Magnetic Fascial Ball
Other: Plantar fascia self massage with a non-magnetic fascia ball — Participants were asked to roll the non-magnetic fascia ball on the sole of each foot for 3 minutes each, from the metatarsal heads towards the heel, concentrating on the medial longitudinal arch. Participants were informed that more intense pressure would be more beneficial and were asked to apply pressure in a way that would not cause pain.
  Arms: Non-Magnetic Fascial Ball

SUMMARY:
In this study, the effect of plantar fascia release with a magnetic fascial cork ball on hamstring and lumbar extensor muscle elasticity will be investigated.

DETAILED DESCRIPTION:
The use of tools such as foam rollers or massage balls to resolve myofascial tension is highly preferred by both therapists and patients. It is theorized that the sweeping pressure generated during rolling causes the fascia to stretch and increase the range of motion. In addition, the warming caused by the friction during rolling can dissolve the adhesions between the fascial layers and restore the elasticity of the myofascial tissues. In addition to similar mechanical effects, the use of cork balls with magnetic properties is becoming increasingly common. Studies have shown that static magnetic magnets reduce pain, increase microcirculation and oxygenation and cause changes in presynaptic membrane function. As far as we know, there is no study examining the myofascial relaxation effect of magnetic balls in the literature. Evaluating the clinical impact and efficacy of this device which allow the person to perform self-massage might contribute the current literature. This study was planned to evaluate the myofascial relaxation caused by two different fascial cork balls with and without magnetic properties.

ELIGIBILITY:
Inclusion Criteria:

* Having scored 3 or less according to the Beighton scoring system
* 18-35 years old,
* Having asymptomatic
* Voluntary participation in the research

Exclusion Criteria:

* Having Beighton score of 4 and above
* Having history of previous surgery
* Having diagnosed pathology of the lower extremities and lumbar region

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Goniometric Measurement of Hamstring Flexibility | Two times in one day (before intervention, immediately after intervention)
  Individuals are positioned supine with the hip of the limb to be measured at 90 degrees. In this position, active knee extension is requested and the acute angle between the long axis of the femur and the long axis of the fibula is measured. The DrGonyometer (iOS) smart phone application, for which a validity and reliability study was conducted, was used for the measurement.

SECONDARY OUTCOMES:
Sit and reach test | Two times in one day (before intervention, immediately after intervention)
  Individuals are placed in a long sitting position with their feet resting on the test battery (Figure 2) and knees in full extension. They are asked to reach forward on the wooden block by placing their hands on top of each other. In this position, the distance between the fingers of the hand and the point where the foot rests is measured and the previous values are recorded as negative and the following values as positive.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Osman PALA, Principal Investigator — Bolu Abant İzzet Baysal Üniversitesi
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No